CLINICAL TRIAL: NCT02215460
Title: Effectiveness of Two Non-surgical Periodontal Treatment Protocols: Randomized Controlled Clinical Trial
Brief Title: Treatment of Periodontitis by Conventional 4 Weekly Sections or Within 24 Hours
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Taubate (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMSQSPT; CEP521/10 (Other: Institutional Ethics Committee on research involving human 521/10); 2010/19079-8 (Other Grant/Funding Number: Fapesp)
Record Dates: First submitted 2014-08-08; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (10):
- Full-mouth scaling (FMS) (Experimental)
  Interventions: Procedure: FMS full-mouth scaling
- FMS chlorhexidine rinse (Experimental)
  Interventions: Procedure: FMS full-mouth scaling; Drug: FMS chlorhexidine rinse
- FMS azithromycin tablets (Experimental)
  Interventions: Procedure: FMS full-mouth scaling; Drug: FMS azithromycin tablets
- FMS placebo rinse (Placebo Comparator)
  Interventions: Procedure: FMS full-mouth scaling; Drug: FMS placebo rinse
- Quadrant scaling (QS) (Experimental)
  Interventions: Procedure: QS quadrant scaling
- QS chlorhexidine rinse (Experimental)
  Interventions: Procedure: QS quadrant scaling; Drug: QS chlorhexidine rinse
- QS azithromycin tablets (Experimental)
  Interventions: Procedure: QS quadrant scaling; Drug: QS azithromycin tablets
- QS placebo tablets (Placebo Comparator)
  Interventions: Procedure: QS quadrant scaling; Drug: QS placebo tablets
- FMS placebo tablets (Placebo Comparator)
  Interventions: Procedure: FMS full-mouth scaling; Drug: FMS placebo tablets
- QS placebo rinse (Placebo Comparator)
  Interventions: Procedure: QS quadrant scaling; Drug: QS placebo rinse

INTERVENTIONS:
Procedure: FMS full-mouth scaling — Participants received oral hygiene instructions and full-mouth scaling within 24 hours. Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: FMS azithromycin tablets; FMS chlorhexidine rinse; FMS placebo rinse; FMS placebo tablets; Full-mouth scaling (FMS)
Procedure: QS quadrant scaling — Participants received oral hygiene instructions and quadrant scaling in 4 weekly sections. Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: QS azithromycin tablets; QS chlorhexidine rinse; QS placebo rinse; QS placebo tablets; Quadrant scaling (QS)
Drug: FMS chlorhexidine rinse — Participants received oral hygiene instructions and full-mouth scaling within 24 hours followed by a 60-day use of 0.12% chlorhexidine mouth rinse (15mL/30 seconds/ 2 times a day). Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: FMS chlorhexidine rinse
Drug: FMS placebo rinse — Participants received oral hygiene instructions and full-mouth scaling within 24 hours followed by a 60-day use of placebo mouth rinse (15mL/30 seconds/ 2 times a day). Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: FMS placebo rinse
Drug: FMS azithromycin tablets — Participants received oral hygiene instructions and full-mouth scaling within 24 hours followed by a 3-day use of azithromycin tablets (1 tablet/day). Debridement procedures were carried out Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: FMS azithromycin tablets
Drug: FMS placebo tablets — Participants received oral hygiene instructions and full-mouth scaling within 24 hours followed by a 3-day use of placebo tablets (1 tablet/day). Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: FMS placebo tablets
Drug: QS azithromycin tablets — Participants received oral hygiene instructions and full-mouth scaling in 4 weekly sections followed by a 3-day use of azithromycin tablets (1 tablet/day). Debridement procedures were carried out Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: QS azithromycin tablets
Drug: QS placebo tablets — Participants received oral hygiene instructions and full-mouth scaling in 4 weekly sections followed by a 3-day use of placebo tablets (1 tablet/day). Debridement procedures were carried out Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: QS placebo tablets
Drug: QS chlorhexidine rinse — Participants received oral hygiene instructions and full-mouth scaling in 4 weekly sections followed by a 60-day use of 0.12% chlorhexidine mouth rinse (15mL/30 seconds/2 times a day). Debridement procedures were carried out Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: QS chlorhexidine rinse
Drug: QS placebo rinse — Participants received oral hygiene instructions and full-mouth scaling in 4 weekly sections followed by a 60-day use of 0.12% placebo mouth rinse (15mL/30 seconds/2 times a day). Debridement procedures were carried out Debridement procedures were carried out under local anesthesia with manual Gracey and McCall curettes and Hirschfield files.
  Arms: QS placebo rinse

SUMMARY:
Periodontitis is a form of gum disease that affects many people in the world. Its traditional protocol of treatment includes oral hygiene instruction and dental scaling to remove debris, dental plaque and tartar in 4 weekly sections. There is an additional time-reduced option also usually cheaper. In this last one, all above described procedures are performed within 24 hours. However, up to now comparative effectiveness between these both types of treatment is not well understood. For, example it is not clear if patients treated in the shorter-time experienced more pain. Therefore, the present study used several parameters to clarify whether beneficial differences between these therapeutic protocols exist or not. In addition, aspects that could help clinicians' and patient's decisions such as experience of pain and anxiety related to dental treatment were also investigated. After receiving verbal and written explanations and signed the informed consent form 150 individuals (n=15/group) having the most common type of periodontitis in adults were randomly allocated to be treated in 4 weekly sections or within 24 hours. Oral hygiene instructions and dental debridement were performed alone or in conjunction with antimicrobial agents: a mouth rinse containing chlorhexidine or systemic azithromycin antibiotic tablets. The parameters measured at baseline, 3, 6 and 9 months after treatment were: indicators of inflammation, amount of oral debris and malodor; quantification of bacteria in plaque samples collected with paper points from teeth and tongue; amount of produced saliva and self-reported questionnaires to collect information about oral condition, daily activities, pain and anxiety related to dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate chronic periodontitis;
* at least 20 natural teeth;
* good general health

Exclusion Criteria:

* systemic diseases or other conditions that could influence the periodontal status;
* events of high blood pressure or diagnosed hypertension;
* alcohol abuse;
* orthodontic devices;
* extended prosthetic fixed devices, removable partial dentures or overhanging restorations;
* pregnancy or breast-feeding;
* history of sensitivity or suspected allergies following the use of oral hygiene products and/or the test antibiotic;
* the need for antibiotic prophylaxis;
* antibiotics and/or anti-inflammatory drug use in the three months prior to the beginning of the study;
* regular use of chemotherapeutic antiplaque/antigingivitis products;
* any furcation lesions;
* periodontal treatment performed within six months prior to study initiation;
* unwillingness to return for follow-up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Improvements in pocket depth and clinical attachment level measurements | Changes in pocket depth and clinical attachment level measurements from baseline to 6 months
  Primary outcomes of effectiveness were improvements of the following clinical parameters: periodontal pocket depth (mm) and clinical attachment level (mm) from baseline to 6 months.

SECONDARY OUTCOMES:
Improvements in plaque index and gingival index | Changes from baseline to 3 months
  Improvements in plaque index (scores) and gingival index (scores) when baseline data was compared to 3 months data.
Maintenance of pocket depth and clinical attachment level measurements | Changes in pocket depth and clinical attachment level from 6 months to 9 months
  Pocket depth (mm) and clinical attachment level (mm) values observed at 6 were compared to those observed at 9 months.
Changes in total bacterial load and levels of selected pathogens | 3 months
  Reductions in total bacterial load and levels of selected pathogens were determined by real time PCR (polymerase chain reaction) in samples from periodontal pockets and dorsal tongue. Values between baseline and 3 months were compared.
Changes in volume of gingival crevicular fluid and levels of pro-inflammatory cytokines | 3 months
  Possible reductions in gingival crevicular fluid volume and in concentrations of tumor necrosis factor alfa (TNFα) and interleukin 1 beta (IL-1β) were measured by comparing values between baseline and 3 months.

OTHER OUTCOMES:
Impact of periodontal treatment on quality of life | 6 and 9 months
  The expected positive effect of periodontal treatment on quality of life (score) was measured by comparing baseline data and data collected at 6 and 9 months after therapy
Impact of periodontal disease on quality of life | Baseline
  The expected negative effect of periodontal disease on quality of life (score) was measured by analyzing baseline data.
Dental Anxiety experience | Baseline
  Dental Anxiety (score) was measured immediately before treatment.
Experience of pain | at the second day for full-mouth scaling groups; or at month for quadrant scaling groups.
  Experience of pain (scale) due to type of scaling was evaluated immediately after treatment.
Changes in nitrite levels | 6 months
  Changes in nitrite levels (mean values) in saliva was determined by comparing baseline and 6 months values.
Improvements in organoleptic and volatile sulphur compounds measurements | 3 months
  The expected positive impact of periodontal treatment on organoleptic (score) and volatile sulphur compounds (mean values) measurements were evaluated at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus of periodontal research of University of Taubate, Taubaté, São Paulo, Brazil

REFERENCES:
- [Result] Cortelli JR, CASTRO MVM; BALEJO RDP, ALENCAR CO, GARGIONI AC, CORTELLI SC, COSTA FO. Clinical and microbiological evaluation of one-stage full-mouth disinfection: a short-term study. Revista de Odontologia da UNESP (Online), v. 42, p. 298-303, 2013. DOI: doi.org/10.1590/S1807-25772013000400010.
- [Result] CORTELLI JR. et al. Clinical/Microbiological Comparative Effects between Full-mouth and Quadrant Debridement plus Chlorhexidine. In: IADR, 2013, SEATTLE. IADR, 2013.
- [Result] CORTELLI JR, COSTA FO, ALENCAR CO, CASTRO MVM, GARGIONI AC, AQUINO DR, CORTELLI SC. CLINICAL EFFECTS OF FULL MOUTH OR QUADRANT DEBRIDEMENT WITH CHLOREXIDINA OR AZITROMYCIN. In: IADR-ASIA PACIFIC REGION, 2013, BANGKOK. IADR-APR, 2013. v. 1. p. 158-158.